CLINICAL TRIAL: NCT01359631
Title: Cephalic Vascular Recording Upon SPG Stimulation in CH Patients - Amendment to the Pathway CH-1 Trial
Brief Title: Cephalic Vascular Recording Upon SPG Stimulation
Status: Completed | Type: Observational
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Henrik Schytz, MD, Human Migraine Research Lab, Dep. Neurology, Glostrup Hospital
Other Study IDs: CIP-001-A
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Cluster Headache
Keywords: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Hypothesis:

Stimulation of the SPG at high frequencies (50-200Hz) is believed to cause a physiological parasympathetic block which decreases VMCA oxyHb concentration and cephalic vessel diameter.

Stimulation of the SPG at low frequencies (1-60 Hz)is believed to cause a physiological parasympathetic upregulation which increases VMCA, oxyHb concentration and cephalic vessel diameter.

DETAILED DESCRIPTION:
Efferent

ELIGIBILITY:
Inclusion Criteria:

•Subject is currently enrolled in Pathway CH-1 (CIP-001)

Exclusion Criteria:

•Subject is NOT currently enrolled in Pathway CH-1(CIP-001)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)